CLINICAL TRIAL: NCT07367529
Title: A Phase Ib/II Clinical Trial to Evaluate the Efficacy and Safety of TQB6411 for Injection in Patients With Advanced Lung Cancer
Brief Title: A Clinical Trial on the Efficacy and Safety of TQB6411 for Injection
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB6411-Ib/II-02
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Advanced Lung Cancer
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB6411 for Injection (Experimental): TQB6411 for Injection is administered every 21 days as a treatment cycle.
  Interventions: Drug: TQB6411 for Injection

INTERVENTIONS:
Drug: TQB6411 for Injection — TQB6411 for Injection is administered every 21 days as a treatment cycle.

SUMMARY:
To evaluate the efficacy and safety of TQB6411 for Injection in subjects with advanced lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study, sign the informed consent form, and demonstrate good compliance;
* Age between 18 and 75 years (calculated based on the date of signing the informed consent form);
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
* Expected survival greater than 12 weeks;
* At least one measurable lesion according to RECIST v1.1 criteria;
* Laboratory test results meeting the following criteria (no blood transfusion within 14 days or hematopoietic growth factor administration within 7 days prior to screening):

  1. Hemoglobin (HGB) ≥ 90 g/L;
  2. Absolute neutrophil count (NEUT) ≥ 1.5×10⁹/L;
  3. Platelet count (PLT) ≥ 90×10⁹/L;
  4. Total bilirubin (TBIL) ≤ 1.5×Upper Limit of Normal (ULN);
  5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN (≤ 5×ULN if liver metastases are present);
  6. Serum creatinine (CR) ≤ 1.3×ULN or creatinine clearance rate (CCR) ≥ 50 mL/min;
  7. Prothrombin time (PT), activated partial thromboplastin time (APTT), and international normalized ratio (INR) ≤ 1.5×ULN (no anticoagulant therapy within the past 2 weeks);
* Lung cancer confirmed by histology or cytology；
* Willing to provide qualified tumor tissue samples for immunohistochemical testing, unless the subject has no eligible archived specimens and is unsuitable or refuses re-biopsy;
* Women of childbearing potential must agree to use effective contraception during the study and for 6 months after study completion, with a negative serum or urine pregnancy test within 7 days before enrollment; male subjects must agree to use effective contraception during the study and for 6 months after study completion (see Section 5.5 for details).

Exclusion Criteria:

* History of or concurrent other malignancies, except for: other malignancies treated with surgery alone and achieving ≥5 years of disease-free survival (DFS); or cured carcinoma in situ of cervix, non-melanoma skin cancer, or superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invading basement membrane)].
* Diseases affecting intravenous injection or blood sampling.
* Adverse reactions from prior therapies not recovered to Common Terminology Criteria for Adverse Events (CTCAE) v6.0 grade ≤1, except for: grade 2 alopecia, grade 2 peripheral neuropathy, grade 2 anemia, non-clinically significant asymptomatic grade 2 laboratory abnormalities, hypothyroidism stabilized with hormone replacement, or other toxicities judged by investigator as non-safety risks.
* Major surgery (Grade 3 or above per National Surgical Classification Catalog 2022), significant traumatic injury within 4 weeks prior to first dose, planned major surgery during study (except protocol-specified procedures), or presence of unhealed wounds/fractures.
* Any bleeding or hemorrhagic events ≥CTCAE grade 3 within 4 weeks prior to first dose.
* Arterial/venous thromboembolic events within 6 months prior to first dose, including: cerebrovascular accidents (including transient ischemic attack (TIA), excluding lacunar infarction), deep vein thrombosis, or pulmonary embolism (implantable venous port- or catheter-related thrombosis or superficial venous thrombosis not considered "severe" thromboembolism).
* Active viral hepatitis with poor control, except: hepatitis B surface antigen (HBsAg)-positive subjects with Hepatitis B virus Deoxyribonucleic acid (HBV DNA) <500 IU/mL (2500 copies/mL) who agree to receive anti-HBV therapy throughout study; or hepatitis C virus (HCV)-infected subjects (Hepatitis C Virus Antibody or Ribonucleic Acid positive) with hepatitis C virus Ribonucleic Acid (HCV RNA) ≤ULN continuing approved antiviral therapy.
* Active syphilis requiring treatment.
* Active tuberculosis, history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced/radiation pneumonitis requiring treatment, clinically significant active pneumonia, history of interstitial lung disease (ILD) requiring treatment, or current ILD.
* History of psychotropic drug abuse or mental disorders.
* Prior or planned allogeneic bone marrow or solid organ transplantation.
* History of hepatic encephalopathy.
* Significant cardiovascular diseases including:

  1. Cardiac dysfunction ≥New York Heart Association (NYHA) class II or Left Ventricular Ejection Fractions (LVEF) <50% by echocardiography;
  2. Clinically significant ventricular arrhythmia history (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes) or arrhythmias requiring continuous antiarrhythmic therapy (subjects with stable atrial fibrillation controlled solely by β-blockers may be included after investigator assessment);
  3. Unstable angina;
  4. Myocardial infarction within 12 months;
  5. Cardio contraction time (QTc) >450ms (male) or >470ms (female) (if abnormal, measure three times at ≥2-minute intervals and average; corrected by Fridericia or Bazett method);
  6. Congenital long QT syndrome or family history.
* Active or uncontrolled severe infection (≥CTCAE grade 2).
* Renal failure requiring hemodialysis or peritoneal dialysis.
* Immunodeficiency including HIV positivity or other acquired/congenital immunodeficiency diseases.
* Uncontrolled autoimmune diseases requiring immunosuppressants or systemic corticosteroids (>10mg prednisone/day equivalent) within 7 days prior to first dose.
* Epilepsy requiring treatment.
* Poorly controlled diabetes (fasting blood glucose >10mmol/L).
* Tumor-related conditions and treatments:

  1. Chemotherapy, immunotherapy, or small-molecule targeted therapy within 3 weeks prior to first dose or within 5 half-lives (whichever shorter); prior local radiotherapy allowed if: completed >4 weeks (>2 weeks for brain) before study treatment, and target lesions are outside radiation field or show progression within field;
  2. National Medical Products Administration (NMPA)-approved traditional Chinese medicines with antitumor indications within 1 week prior to first dose;
  3. Tumor invading major vessels or judged likely to cause fatal hemorrhage;
  4. Uncontrolled effusions/ascites requiring recurrent drainage;
  5. Spinal cord compression, leptomeningeal metastases, or brain metastases with symptoms controlled <4 weeks, or requiring steroids/dehydrating agents within 2 weeks before treatment.
* Known hypersensitivity to study drug or excipients.
* Prior treatment with: Epidermal Growth Factor Receptor/cellular-mesenchymal epithelial transition factor (EGFR/c-Met)-targeted antibody-drug conjugates (ADCs); or topoisomerase I inhibitors (Non-Small Cell Lung Cancer only) or topoisomerase I inhibitor-based ADCs.
* Prior EGFR/c-Met-targeted Monoclonal Antibody (mAbs)/bispecifics with: ≥grade 4 toxicity, permanent discontinuation due to toxicity, ≥grade 3 infusion reactions, or ≥grade 3 myalgia.
* Participation in other antitumor clinical trials within 4 weeks prior to first dose.
* Other conditions judged by investigator to jeopardize subject safety or study completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dosage for the Treatment (RP2D) | Baseline up to 21 days
  Recommended phase II dosage for the treatment of advanced Lung Cancer.
Objective Response Rate (ORR) | Baseline up to 6 mouths
  Objective response rate for the treatment of advanced Lung Cancer.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Baseline up to 6 mouths
  Disease control rate for the treatment of advanced Lung Cancer.
Duration of Relief (DOR) | Baseline up to 2 years
  Duration of relief for the treatment of advanced Lung Cancer.
Progression-Free Survival | Baseline up to 2 years
  Progression-free survival for the treatment of advanced Lung Cancer.
Overall Survival (OS) | Baseline up to 3 years
  Overall survival for the treatment of advanced Lung Cancer.
Adverse Events (AE) | Baseline up to 2 years
  Numbers of participant with incidence and severity of adverse events, serious adverse events, and adverse events associated with investigational drugs (including investigational drugs and control drugs), as well as abnormal laboratory indicators were evaluated.
Incidence of Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (NAb) | Cycle 1 day 1, Cycle 4 day 1, Cycle 6 day 1, Cycle 12 daye 1: 60 minutes before administration (21 days as a treatment cycle)
  Immunogenicity in patients with advanced lung cancer, Incidence of Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (NAb).
Peak concentration (Cmax) | Before administration, 30 minuets, 15 minuets after administration
  The plasma concentration at which the rate of administration and rate of elimination are in equilibrium.
Plasma concentration at steady state (Cav, SS) | Pre-dose of day 1 on multiple dose and 2, 6, 24, 72 hours, 7, 14 days post-dose on multiple dose of day 1
  The plasma concentration at which the rate of administration and rate of elimination are in equilibrium.

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - Beijing Chest Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Affiliated Three Gorges Hospital, Chongqing, Chongqing Municipality
  - The first affiliated hospital of Guangzhou medical university, Guangzhou, Guangdong
  - The first affiliated hospital of Guangzhou medical university, Guanzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Cangzhou Central hospital, Cangzhou, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang People's Hospital, Anyang, Henan
  - Luoyang Central Hospital (Zhengzhou University Affiliated Luoyang Central Hospital), Luoyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjin, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Affiliated Zhongshan Hospital Of dalian University, Dalian, Liaoning
  - Liaoning Cancer Research Institute, Shenyang, Liaoning
  - Shandong First Medical University Affiliated Tumor Hospital, Jinan, Shandong
  - Linyi cancer Hospital, Linyi, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - First Hospital of Shangxi Medical University, Taiyuan, Shangxi
  - Shanxi Cancer hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Air Force Medical University, Xi’an, Shanxi
  - Sichuan cancer hosipital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang